CLINICAL TRIAL: NCT06996756
Title: Gene Therapy for Alpha-1 Antitrypsin Deficiency
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-06027591; 1R61HL169190 (NIH)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: AAT; Emphysema; Gene therapy; DLCO; Augmentation therapy
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- AAV8hAAT(AVL) - 5x10¹¹ gc/kg (Experimental): Lowest dose of vector genome copies per kilogram
  Interventions: Biological: AAV8hAAT(AVL)
- AAV8hAAT(AVL) - 2x10¹² gc/kg (Experimental)
  Interventions: Biological: AAV8hAAT(AVL)
- AAV8hAAT(AVL) - 5x10¹² gc/kg (Experimental)
  Interventions: Biological: AAV8hAAT(AVL)
- AAV8hAAT(AVL) - 2x10¹³ gc/kg (Experimental): Highest dose of vector genome copies per kilogram
  Interventions: Biological: AAV8hAAT(AVL)

INTERVENTIONS:
Biological: AAV8hAAT(AVL) — AAV8hAAT(AVL) gene transfer vector

SUMMARY:
This is a study of gene therapy to treat alpha-1 antitrypsin deficiency. This study aims to treat AAT deficiency with a single administration of AAV8hAAT(AVL), a gene therapy that codes for an oxidation resistant form of the AAT protein, which if safe and if efficacious, will protect the lung on a persistent basis. We hope to learn the safety/toxicity and initial evidence of efficacy of intravenous delivery of this gene therapy to alpha 1-antitrypsin (AAT) deficient individuals.

ELIGIBILITY:
Inclusion Criteria:

* AAT genotype ZZ, or Z null heterozygotes, and if on augmentation therapy, pre-therapy AAT serum levels <11 μM
* Emphysema as assessed by chest high resolution computational tomography (HRCT)
* Lung function parameters consistent with mild to moderate loss of lung function and the presence of emphysema.
* Troponin T within normal limits
* Normal liver ultrasound and serum alpha fetoprotein
* Normal kidney function
* No contraindications to receiving corticosteroid immunosuppression

Exclusion Criteria:

* Individuals receiving systemic corticosteroids or other immunosuppressive medications for pre-existing conditions.
* Inability to tolerate immunosuppression with corticosteroids (e.g., uncontrolled diabetes)
* Individuals with an immunodeficiency disease, or evidence of active infection of any type, including human immunodeficiency virus
* Evidence of major central nervous system, major psychiatric, musculoskeletal or immune disorder
* Prior history of myocardial infarction or cancer within the past 5 years (other than basal cell carcinoma of the skin)
* Decompensated heart failure (NY4A class III-IV at time of baseline clinical assessment)
* Abnormal ECG at screening with findings consistent with cardiac disease
* Females who are currently pregnant or lactating
* Any history of allergies to drugs used for bronchoscopy, including xylocaine, lidocaine, versed, valium, atropine, pilocarpine, isoproterenol, terbutaline, aminophylline, or any local anesthetic
* Individuals receiving experimental medications or participating in another experimental protocol for at least 3 months prior to entry to the study
* Use of oxygen supplementation
* Risk for thromboembolic disease
* History of significant cardiovascular disease, hypertension, prior myocardial infarction and/or cerebrovascular event
* Individuals who are currently on beta-blockers, or other cardiac therapy related drugs
* Prior history of hypersensitivity or anaphylaxis associated with the administration of any AAT product

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety of AAV8hAAT(AVL), as measured by number of subjects with at least 1 serious adverse event. | Approximately 1 year
  Serious adverse events will only be included if assessed as related to the gene therapy.
Toxicity of AAV8AAT(AVL), as measure by number of subjects with any dose limiting toxicity | Approximately 2 years
  If none of the first 4 dosed participants experiences a DLT by the end of Day 28 after treatment (Day 1), the dose of AAV8hAAT(AVL) will be escalated, and the next cohort of participants will start treatment at the next-higher dose level.
Establishing a maximum tolerable dose of AAV8hAAT(AVL) | Approximately 2 years
  If none of the first 4 participants treated at the highest dose level experiences a DLT by the end of Day 28 after treatment, this dose will be determined to be the maximum administered dose (MAD)

SECONDARY OUTCOMES:
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in serum | 4 weeks
  Serum levels of AAT will be measured in the blood
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in serum | 3 months
  Serum levels of AAT will be measured in the blood
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in serum | 6 months
  Serum levels of AAT will be measured in the blood
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in serum | 12 months
  Serum levels of AAT will be measured in the blood
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in serum | 2 years
  Serum levels of AAT will be measured in the blood
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in serum | 3 years
  Serum levels of AAT will be measured in the blood
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in serum | 4 years
  Serum levels of AAT will be measured in the blood
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in serum | 5 years
  Serum levels of AAT will be measured in the blood
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in lung epithelial lining fluid | 12 months
  Levels of AAT in the lung will be measured by bronchoscopy
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in lung epithelial lining fluid | 2 years
  Levels of AAT in the lung will be measured by bronchoscopy
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in lung epithelial lining fluid | 3 years
  Levels of AAT in the lung will be measured by bronchoscopy
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in lung epithelial lining fluid | 4 years
  Levels of AAT in the lung will be measured by bronchoscopy
Efficacy of AAV8hAAT(AVL) as measured by the levels of AAT in lung epithelial lining fluid | 5 years
  Levels of AAT in the lung will be measured by bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- WCMC Department of Genetic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
As the proposed experiments become published in scientific journals, the cleaned, item-level spreadsheet data for all variables will also be shared openly, along with example quantifications and transformations from initial raw data. Final files used to generate specific analyses to answer the Specific Aims and related results will also be shared. The rationale for sharing only cleaned data is to foster ease of data reuse. If any data collection arising from the proposed studies are not shared by publication within one year after the proposed award period ends, the unpublished data will be similarly shared in public domains for ease of access.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the time of publication, and after final analyses have been completed.
Access Criteria: Access to the data may require Material Transfer Agreements, Non-Disclosure Agreements, or other limitations on licensing access and will be managed by the PI